CLINICAL TRIAL: NCT06993779
Title: Whole-slide Image and CT Radiomics Based Deep Learning System for Prognostication Prediction in Upper Tract Urothelial Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Mingzhao Xiao (Other)
Responsible Party: Sponsor-Investigator, Mingzhao Xiao, Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: AI-UTUC; K2024-187-07 (Other: The First Affiliated Hospital of Chongqing Medical University)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: UTUC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AI-UTUC: Patients with Upper Tract Urothelial Carcinoma (UTUC) who underwent radical nephroureterectomy (RNU)
  Interventions: Other: Deep learning system for prognostication prediction in upper tract urothelial carcinoma

INTERVENTIONS:
Other: Deep learning system for prognostication prediction in upper tract urothelial carcinoma — develop and validate a deep learning system for prognostication prediction in upper tract urothelial carcinoma based on CT radiomics and whole slide images.

SUMMARY:
Upper Tract Urothelial Carcinoma (UTUC), characterized by its anatomical complexity and often aggressive clinical behavior, presents substantial difficulties in accurate diagnosis and reliable prognostication. The stratification of postoperative survival utilizing radiomics features derived from imaging and characteristics from whole slide images could prove instrumental in guiding therapeutic decisions to enhance patient outcomes. In this research, our objective is to construct a deep learning-based prognostic-stratification system designed for the automated prediction of overall and cancer-specific survival in individuals diagnosed with UTUC.

DETAILED DESCRIPTION:
Upper Tract Urothelial Carcinoma (UTUC) can be challenging to accurately diagnose and its course difficult to predict, as the disease manifestations and aggressiveness can differ significantly among individuals. This research seeks to create an innovative system employing artificial intelligence to process patient data, encompassing images from diagnostic scans and surgical pathology slides. This system would then be capable of automatically forecasting a patient's overall survival and their specific likelihood of surviving UTUC. Such insights could empower clinicians to tailor more effective treatment strategies for each individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Upper Tract Urothelial Carcinoma (UTUC) who had radical nephroureterectomy (RNU).
* Contrast-enhanced CT scan (e.g., CT urography) less than two weeks before surgery.
* Complete CT image data and clinical data.
* Complete whole slide image data.

Exclusion Criteria:

* Patients with a postoperative diagnosis of non-urothelial carcinoma.
* Poor quality of CT images and/or whole slide image data.
* Incomplete clinical and follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We included patients who had surgery only or who had neoadjuvant chemotherapy before surgery. We excluded patients with a postoperative diagnosis of non-urothelial carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 10 years
  the time from the date of surgery to death from any cause or the date of last contact (censored observation) at the date of data cut-off.

SECONDARY OUTCOMES:
Recurrence free survival | up to 10 years
  the time from the date of surgery to the date of first documented disease recurrence. Patients without recurrence at the time of analysis will be censored

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, The First Affiliated Hospital of Chongqing Medical University, chongqing, chongqing 400016 Recruiting, Chongqing, China

IPD SHARING:
Plan to Share IPD: No
The datasets analyzed during the current study are not publicly available due to the privacy of patients but are available from the corresponding author on reasonable request.